CLINICAL TRIAL: NCT05910450
Title: A 6-month Phase 3, Multicenter, Prospective, Randomized, Double-Blind, Vehicle-Controlled Study, to Evaluate the Efficacy and Safety of Topically Applied Clascoterone Solution for the Treatment of Androgenetic Alopecia in Males, Followed by a 6-month Single-Blind Treatment With Clascoterone or Vehicle Solution
Brief Title: A Study to Evaluate the Efficacy and Safety of Clascoterone Solution in Treatment of Male Pattern Hair Loss
Acronym: SCALP1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cassiopea SpA (Industry)
Collaborators: Ergomed PLC (Network); Pharmapace Inc (Unknown); Canfield Scientific Inc. (Unknown); ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CB-03-01/37
Record Dates: First submitted 2023-06-06; First posted 2023-06-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Alopecia, Androgenetic
Keywords: Alopecia; Androgenetic; Clascoterone solution; Phase 3; Randomized; Double-blind; Vehicle-controlled; AGA
MeSH Terms: conditions — Alopecia | interventions — Clascoterone; Solutions

STUDY DESIGN:
Intervention Model Description: Pivotal, Double-Blind - Part 1: multicenter, prospective, randomized, Double Blind, vehicle-controlled interventional study.
  Extension, Single-Blind - Part 2: subjects who will have completed Pivotal, Double-Blind - Part I of the trial and have been defined as Part 1 responders, will be randomized to be treated, in Single-Blind, for additional 6 months with IMP or vehicle solution.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Clascoterone Part 1 and Part 2 (Experimental): Subjects treated for 12 months with Clascoterone 5% solution (both in double-blind Part 1 and in the single-blind Part 2 of the study)
  Interventions: Drug: Clascoterone 5% solution
- Clascoterone Part 1 + Vehicle Part 2 (Other): Subjects treated for the first 6 months Part 1 in double-blind with Clascoterone 5% solution followed by 6 months Part 2 in the single-blind label with Vehicle
  Interventions: Drug: Clascoterone 5% solution; Drug: Vehicle solution
- Vehicle Part 1 + Clascoterone Part 2 (Other): Subjects treated for the first 6 months Part 1 in double-blind with Vehicle followed by 6 months Part 2 in the single-blind label with Clascoterone 5% solution.
  Interventions: Drug: Clascoterone 5% solution; Drug: Vehicle solution
- Vehicle Part 1 and Part 2 (Placebo Comparator): Subjects treated for 12 months with Vehicle (both in double-blind Part 1 and in the single-blind Part 2 of the study)
  Interventions: Drug: Vehicle solution

INTERVENTIONS:
Drug: Clascoterone 5% solution — Topical application of 1.5 ml of clascoterone solution 5%, twice a day, to balding areas of the scalp (vertex and temples)
  Other Names: CB-03-01 5% solution
  Arms: Clascoterone Part 1 + Vehicle Part 2; Clascoterone Part 1 and Part 2; Vehicle Part 1 + Clascoterone Part 2
Drug: Vehicle solution — Topical application of 1.5 ml of vehicle, twice a day, to balding areas of the scalp (vertex and temples)
  Other Names: Vehicle
  Arms: Clascoterone Part 1 + Vehicle Part 2; Vehicle Part 1 + Clascoterone Part 2; Vehicle Part 1 and Part 2

SUMMARY:
The purpose of the study is to see if Clascoterone can help people with male pattern hair loss to recovery and see if the treatment is effective and safe and how well the drug is tolerated by subjects.

Within this study, the Clascoterone solution will be compared to a placebo.

The study has 2 parts:

Part 1 will see if Clascoterone solution is effective and safe compared to a placebo when applied twice daily for up to 6 months.

Part 2 will see the long-term safety and efficacy of the Clascoterone solution compared to placebo for additional 6 months in subjects defined as ''responders'' in Part 1. A responder is defined as someone who have responded to the study drug, based on research data.

Part 1 of the study is double-blind, meaning that neither the subject nor the study doctor knows which treatment subject is receiving. Part 2 of the study is single-blind and only the study doctor doing the study knows which treatment subject is receiving.

Part 1 of the study will start with baseline visit during which subjects will be randomly assigned (by chance) in ratio 2:1 to apply either Clascoterone or placebo solution to their balding areas of the scalp. Subjects will have 5 clinic visits and 2 follow-up phone calls during 6 months of Part 1 duration. Subjects identified as Part 1 responders at Month 6 visit will be again randomly assigned in ratio 2:1 to receive either study drug or placebo.

Part 2 of the study will consist of 2 additional clinic visits and treatment will last for further 6 months.

Each subject will have also an end of study visit one month after the study drug treatment has been completed or discontinued (it will be one month after end of Part 1 for not responder subjects).

For those subjects who complete the whole study (Part 1 and Part 2), the total duration of the study will be about 14 months, with 12 months of treatment with a total of eight clinic visits and two phone calls.

Subjects taking part in this study will have the medical tests or procedures described below.

* They will be asked about their previous medical history and current medications.
* A brief physical examination will be performed.
* Vital signs, weight and height will be measured.
* Electrocardiograms will be performed.
* Subject's scalp will be checked for any signs of irritation.
* Two different types of photos will be taken during this study: "global photos", i.e. general photos of the subject's scalp and "macro photos", i.e. close up photos of a region of the subject's scalp. Global photos will be taken to help the subject and the study doctor to assess whether there has been a change in subject's hair growth. Macro photos will be used to count the number of hairs in a region of the subject's scalp and measure other properties of the hair (hair width and hair darkness).
* Blood draws and urine sample collection for safety laboratory tests.
* Subject will be asked to complete, on site, the following two questionnaires:

  * Cosmetic Evaluation - a couple of cosmetic questions on acceptability and how easy the study drug is to use.
  * Male Androgenetic Alopecia Questionnaire - some questions about subject's hair assessment.

Eligible subjects will be given a supply of the study drug and shown how to use and store it. The first study drug dose will be applied at the clinic under the supervision of the study staff. Subjects will be instructed to apply about 1.5 ml of study drug with a dropper to the balding areas of the scalp on the vertex and the temples twice daily, once in the morning and once in the evening.

Subjects will be asked to bring back all used containers of study drug and all unused study drug to each study visit. Subjects will also be given a diary, shown what things have to be recorded on it and asked to bring back the completed diary to the study center at each visit.

ELIGIBILITY:
Inclusion Criteria:

Subject can participate in this clinical study if all the following criteria are met:

1. Subject who is male ≥18 years old.
2. Subject who has provided written informed consent.
3. Subject who has mild to moderate AGA in temple and vertex region, rating III vertex to V on the Modified Norwood-Hamilton Scale (i.e., III vertex [IIIv], IV, or V), with a history of ongoing hair loss.
4. Subject who is willing to maintain the same hairstyle, hair length and hair color throughout the study.
5. Subject who is willing to comply with study instructions at home and return to the clinic for required visits.
6. Subject who agrees to continue his shampoo frequency and other general hair care products and regimen for the entire study.
7. Subject who agrees to maintain same dietary and supplement pattern.
8. Subjects who are sexually active with a female partner and are not surgically sterile (vasectomy performed at least 6 months prior to treatment) must agree to use an acceptable form of birth control as described in the informed consent form. For subjects, adequate forms of contraception include condom and spermicide in combination with other forms of female contraception. For females, an acceptable method (Pearl Index <1%) would be to agree to use implants, injectables, combined oral contraceptives, some intrauterine devices, or be postmenopausal (defined as amenorrhea greater than 12 consecutive months in women 50 years of age or older), be surgically sterile (hysterectomy, bilateral tubal ligation [at least 6 months prior], or bilateral oophorectomy).

Exclusion Criteria:

Subjects who meet any of the following criteria are not eligible to participate in the study:

1. Subject who has any dermatological disorders of the scalp in the target region with the possibility of interfering with the application of the IMP or examination method, such as fungal or bacterial infections, seborrheic dermatitis, psoriasis, eczema, folliculitis, scars, or scalp atrophy.
2. Subject who has any skin pathology or condition that, in the investigator's opinion, could interfere with the evaluation of the IMP or requires use of interfering topical, systemic (e.g., uncontrolled thyroid disease, certain genetic disorders that involve hair growth or patterns), or surgical therapy.
3. Subject who has current or recent history (within 6 months) of hair weaves, non-breathable wigs, or hair bonding.
4. Subject who had scalp hair transplants at any time.
5. Subject with a history of active hair loss due to diffuse telogen effluvium, alopecia areata, scarring alopecia, trichotillomania, or conditions/diseases other than AGA.
6. Subject who has a current or recent history (within 6 months) of severe dietary or weight changes or has a history of eating disorder(s), any history of bariatric surgery (gastric bypass, gastric sleeve, stomach stapling); macro- or micro-nutrient deficiencies within the last 6 months (i.e.: clinically significant iron deficiency, protein deficiency confirmed by lab testing) and/or any current diagnosis of malabsorptive disease (i.e.: Celiac, Irritable Bowel disease etc.).
7. Subject who has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this study, including 12-lead electrocardiogram (ECG) findings during the screening period.
8. Subject is currently enrolled in an investigational drug or device study.
9. Subject who has used an investigational drug or investigational device treatment within 30 days or 5 half-lives whichever is longer prior to Visit 2/Baseline.
10. Subject who is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.
11. Subject who has used or is suspected, in the investigator's opinion, to be using anabolic steroids.
12. Subject who may be unreliable for the study, including subjects who engage in excessive alcohol intake or drug abuse, and/or subjects who will be unable to return for scheduled follow-up visits.
13. Subject who has a known hypersensitivity or previous allergic reaction to any of the active or inactive ingredients in the IMPs or tattoo ink.
14. Subject who has used any of the following topical preparations or procedures on the scalp:

    1. Topical scalp treatments for hair growth including minoxidil, Aminexil, hormone therapy, anti-androgens, or other agents that are known to affect hair growth within 12 weeks of Visit 2/Baseline.
    2. Topical scalp over-the-counter (OTC) or cosmetic treatments known or reasonably believed to affect hair growth (e.g., brands such as Maxilene, Nioxin, Foltene, etc.) or hair health or hair growth products with saw palmetto, copper, etc. within 2 weeks of Visit 2/Baseline.
    3. Topical scalp treatments that may have ancillary effect on hair growth including, but not limited to, corticosteroids, pimecrolimus, tacrolimus, and retinoids within 4 weeks of Visit 2/Baseline.
    4. Scalp procedures (surgical, laser, light, or energy treatments, micro-needling, etc.) within 6 months of Visit 2/Baseline.
    5. Platelet rich plasma (PRP) procedure on the scalp within 6 months of Visit 2/Baseline.
15. Subject who has used one or more of the following systemic medications or procedures:

    1. Beta blockers, cimetidine, diazoxide, or corticosteroids (including intramuscular and intralesional injections) within 12 weeks of Visit 2/Baseline. Inhaled, intranasal, or ocular corticosteroids are allowed if use is stable [defined as doses and frequency unchanged for at least 4 weeks prior to Visit 2/Baseline].
    2. Retinoid, isotretinoin, vitamin A intake above 10,000 IU per day, or cyclosporine therapy within 6 months of Visit 2/Baseline.
    3. Any 5 alpha reductase medications (i.e.: Finasteride [Propecia®, etc.], Dutasteride or similar products within 6 months of Visit 2/Baseline.
    4. Chemotherapy or cytotoxic agents at any time.
    5. Radiation of the scalp at any time point.
    6. Other systemic therapy, which in the opinion of the investigator, may materially affect the subject's hair or hair growth, including, but not limited to, spironolactone, vitamin or homeopathy supplement hair growth or hair health products or other steroid hormones (in any form), including anabolic steroids during the 3 months prior to baseline or during the study.
16. Subject who has been previously enrolled in any study with Clascoterone (former CB 03 01).
17. Subject who is an employee or direct relative of an employee of the contract research organization (CRO), the study site, or the Sponsor.
18. Subject who is institutionalized because of legal or regulatory order.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 703 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in non-vellus Total Area Hair Count (TAHC) | 6 months
  Changes from Pivotal Part 1 Baseline in non-vellus Total Area Hair Count (TAHC) at Month 6.
Subject's assessment of own hair coverage | 6 months
  MAA-PRO item 8, a hair coverage-specific PGI-C, as the co-primary endpoint. The clinically meaningful change (threshold) is defined as a response of "1", "2", or "3".
  Note that the item 2 responder threshold was used as a criterion for subjects to qualify for Part 2 enrollment.

SECONDARY OUTCOMES:
Changes in non-vellus TAHC | 3 months
  Changes from Pivotal Part 1 Baseline in non-vellus TAHC at Month 3.
Changes in subject's assessment of satisfaction score | 6 months
  Changes in MAA-PRO SI (Male Androgenetic Alopecia-Patient Reported Outcomes Satisfaction Index) single treatment satisfaction item (item 15) score (i.e. question: "How satisfied are you with the study treatment?") at Month 6, with a minimum value of "Very dissatisfied" and a maximum value of "Very satisfied."

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Mazzetti, M.D., Study Director — Cassiopea SpA
Locations (24):
- United States (16):
  - The Petrus Center for Aesthetic Surgery and Hair Transplantation, North Little Rock, Arkansas
  - Therapeutics Clinical Research, San Diego, California
  - Mayo Clinic, Department of Dermatology, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - DelRicht Research, Baton Rouge, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Henry Ford Health, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - JDR Dermatology Research, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Diane S. Berson MD, PLLC, New York, New York
  - Derm Research Center of New York, Inc., Stony Brook, New York
  - On Site Clinical Solutions, Charlotte, North Carolina
  - DermResearch, Austin, Texas
  - DelRicht Research, Frisco, Texas
  - Progressive Clinical Research, San Antonio, Texas
- Georgia (8):
  - LTD Health, Batumi
  - JSC Curatio, Tbilisi
  - Kanveni National Center of Dermatology and Venerology, Tbilisi
  - Tbilisi Cancer Center, Tbilisi
  - Aversi Clinic, Tbilisi
  - Medi Club, Tbilisi
  - David Abuladze Georgian-Italian Clinic, Tbilisi
  - LTD "Medinvestment", Tbilisi